CLINICAL TRIAL: NCT05656664
Title: Mitigation Efforts in Arsenic Exposure With Folic Acid Supplementation: Reducing Toxicity and Exploring the Impact on Lung Health
Brief Title: Mitigation Efforts in Arsenic Exposure With Folic Acid Supplementation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Kevin Dsouza, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300010144
Record Dates: First submitted 2022-11-10; First posted 2022-12-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Arsenic and/or Arsenic Compound Adverse Reaction
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Study procedures will consist of recruitment of 100 subjects, 50 each in the treatment (Folic Acid, 800 mcg) and placebo groups respectively. Folic Acid 800 mcg or placebo pill bottles will be provided to the participants with instructions to take one pill orally daily. Both the investigators and subjects will be blinded. Compliance will be measured via pill count.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study randomization will be performed by using a randomization scheme provided by the Investigational Drug Service (IDS). The randomization scheme will be held by IDS and concealed to investigators until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo daily 12 weeks
  Interventions: Other: Placebo
- Folic Acid (Experimental): Folic acid 800 ug/day 12 weeks
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Folic Acid — Folic acid supplementation to assess for increased arsenic metabolite excretion
  Arms: Folic Acid
Other: Placebo — Placebo group to assess arsenic metabolite excretion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects on folic acid supplementation in a population living in an environment with chronic arsenic exposure in Birmingham, Alabama.

DETAILED DESCRIPTION:
Folic acid supplementation effects urinary arsenic excretion. In this project investigators propose to investigate if oral folic acid dietary supplementation can increase urinary arsenic metabolite excretion

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Resident of the superfund site
* Clinically stable with no significant changes in general health status in the past 4 weeks prior to screening as assessed by the investigator
* Provide written informed consent

Exclusion Criteria:

* Pregnancy
* Ongoing folic acid nutritional supplementation
* Methotrexate use
* Megaloblastic anemia
* Alcoholic liver disease
* Malabsorptive syndromes - celiac disease, inflammatory bowel disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of urine and blood arsenic metabolites | 12 weeks
  Inorganic As (InAs) within humans undergoes a stepwise biotransformation reaction in which it is methylated to monomethyl-arsonic acid (MMAsIII), and dimethylarsinic acid (DMAsV) facilitating urinary excretion. This occurs via arsenic methyltransferase (AS3MT) using a methyl donor S-adenosylmethionine (SAM). In this pathway the one-carbon unit carried by 5-methyl-tetrahydrofolate (5-MTHF) is transferred to homocysteine to form methionine, which is activated to SAM. Complete methylation to DMAsV is critical as higher proportion of MMAs(III+V) are associated with skin lesions, peripheral vascular disease, atherosclerosis, and cancers.
  We will measure levels of InAs, total DMA and MMA in the urine and blood of the study subjects at baseline and 12 weeks. Outcomes will be reported in percentage (%) of InAs, DMA and MMA in blood and urine.

SECONDARY OUTCOMES:
Respiratory Symptom Questionnaire | 12 weeks
  The Respiratory Symptom Questionnaire (RSQ) is an instrument that assesses the frequency of respiratory symptoms and their impact on patients' activity over the previous four weeks, without requiring a specific diagnostic label of asthma or chronic obstructive pulmonary disease (COPD). The four questions assess the frequency of respiratory symptoms (shortness of breath, wheezing, coughing, and/or chest tightness) during the day and, in response to these respiratory symptoms, frequency of rescue inhaler use, activity limitations and frequency of night-time awakening. We will administer the RSQ to participants at the baseline screening. Maximum value 16, minimum value 4, higher scores represent increased symptom burden.
Pooled Cohort Probability Score | 12 weeks
  The pooled cohort probability score has been used to detect subclinical airway obstruction. Age, sex, race and/or ethnicity, body mass index, smoking status, and smoking pack-years will be obtained and the score will be computed at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Dsouza, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozack AK, Hall MN, Liu X, Ilievski V, Lomax-Luu AM, Parvez F, Siddique AB, Shahriar H, Uddin MN, Islam T, Graziano JH, Gamble MV. Folic acid supplementation enhances arsenic methylation: results from a folic acid and creatine supplementation randomized controlled trial in Bangladesh. Am J Clin Nutr. 2019 Feb 1;109(2):380-391. doi: 10.1093/ajcn/nqy148. PMID 30590411